CLINICAL TRIAL: NCT05053412
Title: Helio Liver Test Case-Controlled Performance Study in China (HEPATIC)
Brief Title: HELIO Liver Test Performance Study in China (HEPATIC)
Acronym: HEPATIC
Status: Completed | Type: Observational
Sponsor: Helio Genomics (Industry)
Collaborators: Helio Health Inc., Irvine, CA (Unknown)
Responsible Party: Sponsor
Other Study IDs: HELIO-2021-CH-001
Record Dates: First submitted 2021-09-16; First posted 2021-09-22 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Hepatocellular Carcinoma and Liver Disease
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- HCC diagnosed Stage 1 (both A and B): 200 stage 1 (A and B) HCC diagnosed patients
  Interventions: Diagnostic Test: Helio Liver Test
- HCC diagnosed Stage 2: 150 stage 2 HCC diagnosed patients
  Interventions: Diagnostic Test: Helio Liver Test
- HCC diagnosed Stage 3: 100 stage 3 HCC diagnosed patients
  Interventions: Diagnostic Test: Helio Liver Test
- HCC diagnosed Stage 4: 50 stage 4 HCC diagnosed patients
  Interventions: Diagnostic Test: Helio Liver Test
- Control liver cancer surveillance subjects: 500 patients total: 250 Subjects with liver cirrhosis, 250 subjects without liver cirrhosis
  Interventions: Diagnostic Test: Helio Liver Test

INTERVENTIONS:
Diagnostic Test: Helio Liver Test — A Helio Liver Test is used as the basis of performance evaluation for specificity and sensitivity for all patients enrolled in the study.

SUMMARY:
De-identified whole blood and serum samples are collected for the purpose of evaluating the performance (sensitivity/specificity) of the HelioLiver Test for the detection of hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
The purpose of this study is to define the performance characteristics (sensitivity and specificity) of the Helio Liver Test within a study population of subjects that have been diagnosed with liver cancer at various stages (I to IV) and for control subjects who have been confirmed to not have liver cancer by at least one imaging technique, such as ultrasound, MRI or CT. Control subjects will include patients who are at high-risk for liver cancer and have been recommended to undergo liver cancer surveillance.

ELIGIBILITY:
Inclusion Criteria:

* The subject has provided informed consent to participate in the study
* The subject is 18 to 75 years old (inclusive)

For subjects diagnosed with HCC, the subject must meet the following criteria:

* The subject must have active HCC at the time of the blood draw
* The subject has not undergone treatment for HCC

For subjects diagnosed with primary liver cancer, the subject has been recently diagnosed (within 3 months of enrollment) to have HCC by at least one of the following methods:

* Subject has a ≥1 cm lesion that is indicated to be HCC by MRI or CT due to exhibiting arterial phase hyperenhancement in combination with washout appearance
* Subject has a lesion of any size that is indicated to be HCC due to capsule appearance by 4 phase CT scan or multiphase contrast enhanced MRI
* Subject has a biopsy that is positive for HCC
* Diagnostic imaging by multiphasic MRI or CT indicates a suspicious lesion on the liver, which is subsequently confirmed to be HCC by another method (biopsy, or surgical pathology) within 3 months from the blood draw

For subjects without liver cancer, the subject is confirmed NOT to have liver cancer by at least one of the following methods within 3 months of the blood draw

* Ultrasound result is negative for HCC or suspicious lesions
* Diagnostic imaging by multiphasic MRI or CT clearly indicates the subject does not have HCC

Exclusion Criteria:

* Subject has previously been diagnosed with a primary liver cancer

  * Subject has previously received any treatment for HCC prior to enrollment/blood sample collection, including: surgery, ablation, embolization, pharmacotherapy, radiotherapy, liver transplant or other treatment indicated for HCC
  * Subject has undergone prior or current treatment for HCC with sorafenib, regorafenib, or other treatment indicated for HCC.
  * Subject has received a cancer diagnosis within the past 5 years for any cancer (with the exceptions of basal cell or squamous cell skin cancers).
  * Subject has received treatment for any cancer, including chemotherapy and/or radiation therapy, within 5 years prior to enrollment/sample collection.
  * Subject have received IV contrast dye (for multiphasic CT or MRI) within 1 day [or 24 hours] of blood collection.
  * Subject has undergone fine needle aspiration (FNA) of target pathology withing 3 days prior to blood collection.
  * Subject has undergone a biopsy (other than FNA) of target pathology withing 7 days prior to blood collection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have been clinically diagnosed with HCC, or are negative for HCC after regular surveillance will be enrolled. Approximately 1,000 subjects total will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 1556 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
evaluate sensitivity and specificity of Helio Liver Test | enrollment period
  To evaluate the performance characteristics (sensitivity and specificity) of the Helio Liver Test within a population of subjects diagnosed with HCC or Control Subjects who are at high-risk of HCC due to a benign liver condition.

SECONDARY OUTCOMES:
secondary subset analysis for sensitivity | enrollment period
  The sensitivity of the Helio Liver Test will be calculated based on cancer stage
secondary subset analysis for sensitivity and specificity | enrollment period
  The sensitivity and specificity of the Helio Liver Test will be evaluated based upon the underlying cause of liver cirrhosis
secondary subset for sensitivity and specificity by severity of liver cirrhosis | enrollment period
  Sensitivity and specificity by severity of liver cirrhosis (Child-Pugh score)

CONTACTS AND LOCATIONS:
Overall Officials: RIchard Van Etten, MD, PhD, Study Chair — University of California, Irvine
Locations (2):
- China (2):
  - People's Liberation Army General Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guangzhou Medical University, Beijing

IPD SHARING:
Plan to Share IPD: Undecided